CLINICAL TRIAL: NCT00295074
Title: The Effect of Mild Traumatic Brain Injury on Recovery From Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0402095
Record Dates: First submitted 2006-02-17; First posted 2006-02-22 (Estimated); Last update posted 2008-02-11 (Estimated); Status verified 2008-02

CONDITIONS: Traumatic Brain Injury; Trauma; Head Injury; Brain Concussion
Keywords: traumatic brain injury; head injury; concussion; neuropsychologic test
MeSH Terms: conditions — Brain Injuries, Traumatic; Wounds and Injuries; Craniocerebral Trauma; Brain Concussion | interventions — Neuropsychological Tests

INTERVENTIONS:
Procedure: neuropsychologic testing

SUMMARY:
Mild traumatic brain injury (TBI) is a common injury that can produce significant functional sequelae and ongoing disabling symptoms. Predicting who will have an uncomplicated recovery and who will suffer ongoing symptoms is difficult. This protocol evaluates the use of neuropsychologic testing after mild TBI in injured patients to attempt to objectively establish predictors of long term disability and functional recovery.

DETAILED DESCRIPTION:
Patients who are hospitalized and who have suffered mild TBI (loss of consciousness or post-traumatic amnesia; Glasgow Coma Score 13-15; admitted within 24 hours of injury; able to read, speak, and understand English) who do not have pre-injury dementia or significant cognitive impairment will undergo computerized neuropsychologic testing using a previously validated tool that has been effective in sports-related mild TBI. Sequential testing will be performed during recovery and patients who report disabling symptoms and/or functional impairment will be compared to patients who recover uneventfully. Goal is to identify those parameters that predict early who may suffer long term sequelae or functional impairment and therefore benefit from early cognitive rehabilitation. Secondary goals are to establish objective parameters for functional recovery after mild TBI.

ELIGIBILITY:
Inclusion Criteria:

* Mild TBI
* Admitted within 24 hours of injury
* Able to read, speak,and understand English

Exclusion Criteria:

* Expected to die of their injuries
* Pre-existing dementia or significant cognitive impairment
* Neurologically impaired and incapable of completing testing
* Physically incapable of using arms/hands to complete computerized testing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2004-10; Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
functional outcome
subjective symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Brian G Harbrecht, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center-Presbyterian, Pittsburgh, Pennsylvania, United States